CLINICAL TRIAL: NCT03685617
Title: Comparsion of the Effects of the Histobal Pacing and Double-lumen Pacing on the Function of Left Atrium in Short Term
Brief Title: Effect of His Bundle Pacing in Treatment of Slow Arrhythmia on Function of Left Atrial and Ventricle in Short Term
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Ruiqin xie, Director of the Department of Cardiology in the Second Hospital of Hebei Medical University, The Second Hospital of Hebei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XieRuiqindoctorHBP
Record Dates: First submitted 2018-08-25; First posted 2018-09-26 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Slow Arrhythmia; His Bundle Pacing; Function of Left Atrial and Ventricle

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Dual chamber pacemaker (Active Comparator): 1. Patients with sinus node disfunction: sinus node disfunction with obvious clinical symptoms, including sinus pause; patients with chronotropismus disfunction; patients have to take some medicine due to some diseases, but the medicine may result to sinus bradycardia.
  2. Adult Acquired Atrioventricular Block (AVB): (1). Third degree or advanced atrioventricular block in any block part with symptomatic bradycardia (2). Patients taking other antiarrhythmic drugs in long term, which could result in third degree or advanced AVB (in any block part) and symptomatic bradycardia;
  3. Patients with acute myocardial infarction (AMI) and AVB:
  (1). Patients with His-Purkinje system persistent second degree AVB and retardant or third degree AVB after STEMI; (2). Patients with temporary severe second degree AVB or third degree AVB (block part under atrioventricular node) and retardant; 4. Patients with carotid sinus hypersensitivity or neurogenic syncope of the heart;
  Interventions: Device: Dual Chamber Pacemaker
- His bundle pacemaker (Experimental): His Bundle Pacemaker: All of the Criteria Inclusion of dual chamber pacemaker excluding patients with block part under the his bundle;
  Interventions: Device: His Bundle Pacemaker

INTERVENTIONS:
Device: Dual Chamber Pacemaker — 1. Conducting venipuncture. Subclavian vein is our first choice. Then we set up two venous channels and implant two guiding wires into postcava. 2.Putting 2 sheathing canals into heart along with guiding wires. 3.Locating the sheathing canals, and putting electrodes into canals. 3.Adjusting the electrodes and revolving them anticlockwise to lead them to right atrium and right ventricle respectively under the X-ray. 4.Immobilizing electrodes. 5. Some ways to determine whether the electrode is fixed or not: the head of the electrodes could beat rhythmically with atrium or ventricle or by testing damage current. 6.Removing the canals and suturing.
  Arms: Dual chamber pacemaker
Device: His Bundle Pacemaker — 1.Conducting venipuncture. Subclavian vein is our first choice. Then we set up two venous channels and implant two guiding wires into postcava. One of the guide wire is 120cm in length, 0.035 or 0.038 in diameter, which is required to lead the C315 sheathing canal. 2.Putting C315 sheathing canal into heart along with guiding wires. 3.Locating the C315 sheathing canal, and adjusting the head of C315 towards ideal pacing location. 3.Implanting the spiral electrodes and fixing them. Leading the spiral electrode to the side of his bundle along the C315 canal under the X-ray. The other electrode is leaded to right atrium like dual chamber pacemaker under the X-ray. 4.Revolving the 3830 electrode suitably to Immobilizing it in cardiac muscle. If the electrode can get his electric potential and produce his bundle pacing successfully, we revolve the 3830 electrode and immobilize it.
  Arms: His bundle pacemaker

SUMMARY:
Bradyarrhythmia is one of the common diseases. Also, bradyarrhythmia could result in syncope, clinic convulsion, shock, sudden death and so on, which could influence people's life quality severely. Artificial pacemaker is the only way that can cure bradyarrhythmia. However, traditional right ventricular apical pacing, because its electric stimulation is mostly different of the physiological one, could lead to ventricular thick inhomogeneously. At the same time, traditional right ventricular apical pacing also could result in cardiac arrhythmia and fibrosis, dyssynchrony of the ventricles, which can increase the volume of mitral regurgitation. Besides, cardiac resynchronization therapy (CRT), which aims to cure chronic heart failure, is also unsatisfactory. On the contrary, the electric stimulation of his bundle pacing (HBP) is the same as the physiological one, which produces a relatively normal electrical stimulation and synchrony in systolic velocities in ventricular. Thus, HBP could produce a better haemodynamic effect, which is the hotspot in pace-making area recently.

The purpose of this study is to conduct a comparison in patients' cardiac function, ECG, and pacemakers' threshold value, time limit and so on among dual chamber pacemaker and HBP.

DETAILED DESCRIPTION:
The purpose of this study is to conduct a comparison in patients' cardiac function, ECG, and pacemakers' threshold value, time limit and so on among dual chamber pacemaker and HBP.

The clinic trial is about to conduct pacemaker implantation in 84 participants, which distribute into dual chamber pacemaker, HBP 2 groups in proportion of 1:1 in random. All of the participants are supposed to conduct ultrasonic cardiogram (UCG), ECG, BNP and pacemaker programing.

Methods: conduct pacemaker implantation in 84 patients, which distribute into dual chamber pacemaker, HBP 2 groups in proportion of 1:1 in random. Patients with The implanting progress of dual chamber pacemaker: 1. Conducting venipuncture. Subclavian vein is our first choice. Then investigator will set up two venous channels and implant two guiding wires into postcava. 2.Putting 2 sheathing canals into heart along with guiding wires. 3.Locating the sheathing canals, and putting electrodes into canals. 3.Adjusting the electrodes and revolving them anticlockwise to lead them to right atrium and right ventricle respectively under the X-ray. 4.Immobilizing electrodes. 5. Some ways to determine whether the electrode is fixed or not: the head of the electrodes could beat rhythmically with atrium or ventricle or by testing damage current. 6.Removing the canals and suturing.

The implanting progress of HBP: 1. Conducting venipuncture. Subclavian vein is our first choice. Then investigator will set up two venous channels and implant two guiding wires into postcava. One of the guide wire is 120cm in length, 0.035 or 0.038 in diameter, which is required to lead the C315 sheathing canal. 2.Putting C315 sheathing canal into heart along with guiding wires. 3.Locating the C315 sheathing canal, and adjusting the head of C315 towards ideal pacing location. 3.Implanting the spiral electrodes and fixing them. Leading the spiral electrode (type 3830 on Medtronic) to the side of his bundle along the C315 canal under the X-ray. The other electrode is leaded to right atrium like dual chamber pacemaker under the X-ray. 4.Revolving the 3830 electrode suitably to Immobilizing it in cardiac muscle. If the electrode can get the his electric potential and produce his bundle pacing successfully, investigator revolve the 3830 electrode and immobilize it. 5. Some ways to determine whether the electrode is fixed or not: the head of the electrodes could beat rhythmically with atrium or ventricle or by testing damage current. 6.Removing the canals and suturing.

Both of the dual chamber pacemaker and the HBP should ensure to keep 100% pacemaking rate in 60-70 bpm heart rate.

All of the participants are supposed to be tested ECG, UCG and some pacemaker programming on pre-operation and 7 days after the operation.

Collection of relevant data:

Threshold value, sense and damage current of pacemaker. Two technologists of the pacemaker detect the threshold value, sense and damage current of the pacemakers respectively. Then all the data will be collected in average value.

UCG: testing the sizes of left atrium (LA), right atrium (RA), left ventricle (LV), right ventricle (RV) before and after the operation. Besides, the ejection fraction (EF) of LV and LA, and E peak, A peak and velocity time integral (VTI) of LA will be tested during the examination. All of the examination will be completed by one cardiologist and one physician of cardiac uhrasonography. Meanwhile, patients should complete BNP testing during the follow-up visit pre-operation and 7 days after the operation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with sinus node disfunction: sinus node disfunction with obvious clinical symptoms, including sinus pause; patients with chronotropismus disfunction; patients have to take some medicine due to some diseases, but the medicine may result to sinus bradycardia.
2. Adult Acquired Atrioventricular Block (AVB):

2.1.Third degree or advanced atrioventricular block in any block part with symptomatic bradycardia

2.2.Patients taking other antiarrhythmic drugs in long term, which could result in third degree or advanced AVB (in any block part) and symptomatic bradycardia;

2.3.Patients with carotid sinus hypersensitivity or neurogenic syncope of the heart;

Exclusion Criteria:

1.Patients with congenital heart diseases,such as arial septal defect,ventricuar defect, rheumatic heart diseases, and valvular heart diseases,such as MS, MI, TS, TI.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Changes of ECG | baseline,1 and 7 days after the operation
  time limit of QRS in ms, PR duration in ms, QRS duration and QT duration in ms
Changes of the Data of Pacemaker | 1 and 7 days after the operation
  Threshold value in V, sense in mV of the pacemaker
Changes of UCG | baseline,1 and 7 days after the operation
  UCG:sizes of LA,RA,LV,RV in mm, and ejetion fraction of LV and LA (%), and E peak, A peak in mm and velocity time integral (VTI) of LA
Changes in BNP | baseline,1 and 7 days after the operation
  BNP in pg/ml

CONTACTS AND LOCATIONS:
Locations (1):
- Second Hospital of Hebei Medical University, Shijiazhuang, Hebei, China